CLINICAL TRIAL: NCT04215562
Title: Outcome and Complications of Peripheral Facial Palsy Following Rehabilitation: A Retrospective Study
Brief Title: Outcome of Facial Palsy Following Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Yousra Hisham Abdel Fattah, Lecturer of Physical Medicine, Rheumatology and Rehabilitation, University of Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 0304299
Record Dates: First submitted 2019-12-29; First posted 2020-01-02 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-05

CONDITIONS: Facial Paralysis
MeSH Terms: conditions — Facial Paralysis | interventions — Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with peripheral facial palsy (Other): collection of data from records on the outcome of rehabilitation therapy on patients with peripheral facial palsy and types of complications associated with this therapy type
  Interventions: Combination Product: rehabilitation

INTERVENTIONS:
Combination Product: rehabilitation — electro-therapy, heat therapy, massage and exercise therapy

SUMMARY:
Retrospective case series,the aim of this study is to assess the outcome and rate of complications in patients with facial palsy following rehabilitation, a retrospective study.

DETAILED DESCRIPTION:
Data from all patients presenting to the outpatient clinics of the Physical Medicine, Rheumatology and Rehabilitation Department. Faculty of Medicine, Alexandria University in the past 3 years will be collected. The outcome and complications from rehabilitation of facial palsy will be recorded.

Primary Outcome: complications of Facial palsy following rehabilitation. Confidentiality of all records will be ensured.

ELIGIBILITY:
Inclusion Criteria:

* all patients with primary idiopathic peripheral facial palsy

Exclusion Criteria:

* all patients with secondary causes of facial palsy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
prognosis or outcome of therapy | 3-6 months
  have patients recovered fully, partially or did not recover
complications | 3-6 months
  types of complications developed during rehabilitation

CONTACTS AND LOCATIONS:
Overall Officials: Yousra Hisham A Fattah, Principal Investigator — Alexandria University Faculty of Medicine
Locations (1):
- Alexandria University, Faculty of Medicine, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No